CLINICAL TRIAL: NCT04115709
Title: Decision Support System to Evaluate VENTilation in ARDS (DeVENT)
Brief Title: Decision Support System to Evaluate VENTilation in ARDS
Acronym: DeVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: European Commission (Other); Mermaid A/C (Unknown); Aalborg University (Other); Université d'Auvergne (Other); Medical University of Vienna (Other); Sorbonne University (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19IC5421
Record Dates: First submitted 2019-09-02; First posted 2019-10-04 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Intensive Care; Device; Beacon Caresystem©; Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Device attached with advice activated (Experimental): Beacon Caresystem device will be attached to the patients and its ventilator advice will be activated.
  Interventions: Device: Beacon Caresystem device with advice
- Control: standard care with device attached without advice (Active Comparator): Beacon Caresystem device will be attached to the patients however the ventilator advice will be deactivated.
  Interventions: Device: Beacon Caresystem device without advice activated

INTERVENTIONS:
Device: Beacon Caresystem device with advice — Beacon Caresystem device provides ventilator settings advice to Doctors
  Arms: Intervention: Device attached with advice activated
Device: Beacon Caresystem device without advice activated — Beacon Caresystem device does not give ventilator settings advice
  Arms: Control: standard care with device attached without advice

SUMMARY:
Patients with Acute Respiratory Distress Syndrome (ARDS) residing in the intensive care unit (ICU) often require support for their breathing from a mechanical ventilator to provide adequate gas exchange, and although it is life-saving in this setting, it is also known to contribute to the morbidity and mortality in the condition.

Mechanical ventilation delivers a volume and pressure of gas for each breath and can vary oxygen levels. Selecting the correct oxygen, pressure and volume levels is important, as incorrect levels can harm the patient, and result in an increased time connected to the ventilator.

Recently, a system has been developed (the Beacon Caresystem) which advises the healthcare practitioner by the bedside as to how to best set the ventilator. This system is based on mathematics which describes the patients disease and may therefore provide ventilator settings which better suit the individual.

The purpose of this study is to compare mechanical ventilation in ARDS patients following advice from the Beacon Caresystem to that of standard care to investigate whether the use of the system results in improved ventilation in all severities and phases of ARDS and thus reducing morbidity in ARDS. The investigators plan to recruit 110 patients (50 in the UK and 30 in each of the other 2 sites). The study also aims to examine the biological and physiological factors that determine the worsening of ARDS and the processes involved in recovery from ARDS with the aim to develop new therapies to help detect the condition and improve recovery.

The investigators will utilise all raw data will be collected from the Beacon Caresystem to physiologically characterise the progression and resolution phases of ARDS.

Additionally blood and Urine samples will be taken from healthy volunteers (100 in total) as a control comparison group for the biological analyses carried out in the DeVENT study.

DETAILED DESCRIPTION:
The study is a randomised control trial, comparing the effects of mechanical ventilation in ARDS provided as standard care, with mechanical ventilation set according to the advice of the Beacon Care system. The study will compare if the use of the system results in a better application of PEEP and driving pressure across all severities and phases of ARDS.

The broad timeframe for the study is as follows. The study will be conducted at three sites. Two of these sites are outside the UK, one in France and one in Italy.

The systems will be delivered and installed starting September/October 2019 in the UK site, followed by France and Austria in November 2019. A one month period of training will then follow where all doctors and nurses involved in using the system will be trained. During this period none of the systems advice will be applied. This training will be supported by study partners, and nurses trained as super users of the system, by Mermaid Care A/S, the company producing the system, and by project investigators who have previously conducted studies using the system.

Patient inclusion and data collection will be performed at in the UK sites over a 15 month period from start October 2019 to January 2020. In both European sites, inclusion and data collection will be performed over a 12 month period from start January 2020 to December 2020. Final data analysis and report writing will be performed by March 2021.

For all study sites, all adult patients diagnosed with ARDS in the cardio-thoracic intensive care unit (ICU) undergoing mechanical ventilation will be considered to see if they are eligible for the study.

Patients will only be considered eligible if they are Within 7 days of an acute and potentially reversible episode of acute respiratory failure, their chest radiograph with bilateral infiltrates is consistent with evidence of pulmonary oedema but not fully explained by cardiac failure and they present with hypoxaemia. In addition, patients are not considered eligible due to being aged under 18, not having an arterial catheter for blood sampling at study start, consent declined, over 7 days of mechanical ventilation, treatment withdrawal imminent within 24 hours, Do Not Attempt Resuscitation order in place and for having a severe chronic respiratory disease requiring domiciliary ventilatioin. For each patient, if identified as eligible, advice to participate in the study will be sought.

Critically ill patients are and often unconscious and may not be able to grant consent. Therefore, the Patient Informed Sheet (PIS) and Consent Form will be requested from a third party acting as a consultee; in most cases this person will be a Personal Consultee, who is someone who knows the person lacking capacity and is able to advise the researcher about that person's wishes and feelings in relation to the project and whether they should join the research. This person must be interested in the welfare of the patient in a personal capacity, not in a professional capacity or for remuneration and will mostly likely be family member, carer or friend, etc. Where the personal consultee is not available on site, the researcher may contact the personal consultee by telephone and seek verbal advice. The verbal agreement will be recorded in the telephone consultee declaration form. The telephone consultee declaration form will be signed by a second member of staff who has witnessed the telephone advice. A copy of the PIS will be emailed to the personal consultee.

Where no Personal Consultee is available, the researcher will nominate a professional person to assist in determining the participation of a person who lacks capacity. A Nominated Professional Consultee is someone who will be appointed by the researcher to advise the researcher about the person's (who lacks capacity) wishes and feelings in relation to the project and whether they should join the research. An independent clinician not treating the patient will be asked to be the nominated consultee. A patient information sheet will be distributed immediately following the patient being identified as eligible for the study.

The study investigators will ask the patient if they can use their existing hospital records. Without their consent, no additional information about the patient will be collected for the purposes of the study. However, to maintain integrity of the randomised trial, all information collected up to that time will still be used and analysed as part of the study.

If consent is obtained and the patient is still eligible, then they will be randomly allocated to one of two groups. This random allocation will be performed according to the randomisation template with random block allocation.

If the patient is allocated to the standard care group then all care will be according to usual practice. If the patient is allocated to the Beacon group, mechanical ventilation will be set with advice from the system. In either case, the study ends for the individual patient either with successful transfer of the patient to another department, or patient death. All other care will be according to usual practice.

110 patients will be included in the study, with 55 patients in each of the groups. 55 patients per group will allow to detect a difference of 3cmH2O in driving pressure between the groups with 90% power and a two sided alpha of 0.05 assuming a control group driving pressure of 15 cmH2O with a standard deviation of 2.5 cmH2O and including a 40% dropout. The investigators have used data from the MIMIC dataset (as published in Serpo Neto et al) for the estimation of the driving pressure. In view of the longitudinal analysis, loss to follow up has taken account of an average mortality of 34% and a 6% drop out.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation.
* Within 1 week of a known clinical insult or new or worsening respiratory symptoms
* Chest radiograph with bilateral infiltrates consistent with evidence of pulmonary oedema but not fully explained by cardiac failure.
* Hypoxaemia as defined by PaO2/FiO2 of ≤ 300mmHg (or ≤ 40kPa) (pre-ECMO PaO2/FiO2 will be used should patient be placed on extracorporeal support).

Exclusion Criteria:

* Age < 18 years old.
* The absence of an arterial catheter for blood sampling at study start.
* Consent declined.
* Over 7 days of mechanical ventilation.
* Treatment withdrawal imminent within 24 hours.
* DNAR (Do Not Attempt Resuscitation) order in place
* Severe chronic respiratory disease requiring domiciliary ventilation (except for sleep disordered breathing)
* Veno-Arterial ECMO

Healthy Volunteer Sample collection:

Inclusion Criteria

* 18 years or older
* Able to consent
* Have mental capacity

Exclusion Criteria

* Blood borne viruses: HIV, Hep B, Hep C
* Blood taken in the last 7 days
* Under doctor for investigation
* Haematological disease
* Currently suffers from infection
* Needle phobia
* Problems with veins / vessels
* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Average Driving pressure delivery by the mechanical ventilator | 18 months
  To assess the average driving pressure delivered by the mechanical ventilator over the period of time when ARDS ventilation management is advised by the Beacon Caresystem as compared to standard care.

SECONDARY OUTCOMES:
Daily Average physiological status - oxygenation (SpO2) | 18 months
  • Daily average physiological status defined as daily averages of measured values of oxygenation (SpO2)
Daily Average physiological status - end-tidal CO2 fraction (FE'CO2) | 18 months
  • Daily average physiological status defined as daily averages of measured values end-tidal CO2 fraction (FE'CO2)
Daily Average physiological status - metabolism (VO2, VCO2) | 18 months
  • Daily average physiological status defined as daily averages of measured values of metabolism (VO2, VCO2)
Daily Average physiological status - ventilation (respiratory rate) | 18 months
  • Daily average physiological status defined as daily averages of measured values of ventilation (respiratory rate)
Daily Average physiological status - ventilation (tidal volume) | 18 months
  • Daily average physiological status defined as daily averages of measured values of ventilation (tidal volume)
Daily Average physiological status - ventilation (anatomical dead space) | 18 months
  • Daily average physiological status defined as daily averages of measured values of ventilation (anatomical dead space)
Daily Average physiological status - pulmonary mechanisms (mean airway pressure) | 18 months
  • Daily average physiological status defined as daily averages of measured values of pulmonary mechanisms (mean airway pressure)
Daily Average physiological status | 18 months
  • Daily average physiological status defined as daily averages of measured values of pulmonary mechanisms (respiratory system compilance)
Daily Average physiological status | 18 months
  • Daily average physiological status defined as daily averages of measured values of ventilator settings
Daily Average physiological status - PaO2/FiO2 | 18 months
  • Daily average physiological status defined as daily averages of measured values of PaO2/FiO2
Daily Average physiological status - shunt fraction | 18 months
  • Daily average physiological status defined as daily averages of measured values of shunt fraction
Daily Average physiological status - end-expiratory lung volume | 18 months
  • Daily average physiological status defined as daily averages of measured values of end-expiratory lung volume over time as continuously measured by the Beacon system
Daily average calculated delivered pressure over time | 18 months
  • Daily average calculated delivered pressure over time, for periods of spontaneous breathing.
Daily average calculated mechanical power over time | 18 months
  • Daily average calculated mechanical power over time
Daily average calculated oxygenation index over time | 18 months
  • Daily average calculated oxygenation index over time
Daily average ventilatory ratio over time | 18 months
  • Daily average ventilatory ratio over time
Incidence and duration of proning events and pre- and post- respiratory physiology | 18 months
  • Incidence and duration of proning events and pre- and post- respiratory physiology
Ventilator free days at 28 days. | 28 days
  • Ventilator free days at 28 days.
Composite endpoint including any cause of death at 28 days and days free of mechanical ventilation within 28 days among survivors | 28 days
  • Composite endpoint including any cause of death at 28 days and days free of mechanical ventilation within 28 days among survivors
Time from control mode to support mode | 18 months
  • Time from control mode to support mode
Proportion of breaths dysyncronous with the ventilator | 18 months
  • Proportion of breaths dysyncronous with the ventilator
Number of changes in ventilator settings per day | 18 months
  • Number of changes in ventilator settings per day
Percentage of time in control mode ventilation | 18 months
  • % of time in control mode ventilation
Percentage of time in support mode ventilation | 18 months
  • % of time in support mode ventilation
Total duration of mechanical ventilation | 18 months
  • Total duration of mechanical ventilation
Changes in tidal volume over time | 18 months
  • Changes in tidal volume over time
Changes in Positive End Expiratory Pressure (PEEP) setting over time | 18 months
  • Changes in Positive End Expiratory Pressure (PEEP) setting over time
Daily and cumulative fluid balance. | 18 months
  • Daily and cumulative fluid balance.
Timing, incidence and duration of ECMO | 18 months
  • Timing, incidence and duration of ECMO
Timing, incidence and duration of neuromuscular blockade | 18 months
  • Timing, incidence and duration of neuromuscular blockade
Mortality at 28 days | 28 days
  Mortality at 28 days
Mortality at 6 months | 6 months
  Mortality at 6 months
Mortality at 1 year | 1 year
  Mortality at 1 year
Organ failure assessment (SOFA) score and/or delta SOFA | 28 days
  • Organ failure free days in the first 28 days, assessed using the sequential organ failure assessment (SOFA) score and/or delta SOFA
Number of patients with ventilation related complications | 18 months
  Number of patients with ventilation related complications e.g. pneumothorax and/or pneumomediastinum
Device malfunction event rate | 18 months
  • Device malfunction event rate
Number of times the advice from the Beacon system is followed | 18 months
  • Number of times the advice from the Beacon system is followed

CONTACTS AND LOCATIONS:
Overall Officials: Brijesh Patel, MBBS MRCP FRCA FFICM PhD, Principal Investigator — Imperial College London
Locations (3):
- Medical University of Vienna, Vienna, Waehringer Guertel, Austria
- Université Clermont Auvergne, Clermont-Ferrand, France
- Imperial College London, Royal Brompton Hospital campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel BV, Mumby S, Johnson N, Handslip R, Patel S, Lee T, Andersen MS, Falaschetti E, Adcock IM, McAuley DF, Takata M, Staudinger T, Karbing DS, Jabaudon M, Schellongowski P, Rees SE; DeVENT Study Group. A randomized control trial evaluating the advice of a physiological-model/digital twin-based decision support system on mechanical ventilation in patients with acute respiratory distress syndrome. Front Med (Lausanne). 2024 Oct 30;11:1473629. doi: 10.3389/fmed.2024.1473629. eCollection 2024. PMID 39540041
- [Derived] Patel B, Mumby S, Johnson N, Falaschetti E, Hansen J, Adcock I, McAuley D, Takata M, Karbing DS, Jabaudon M, Schellengowski P, Rees SE; DeVENT study group. Decision support system to evaluate ventilation in the acute respiratory distress syndrome (DeVENT study)-trial protocol. Trials. 2022 Jan 17;23(1):47. doi: 10.1186/s13063-021-05967-2. PMID 35039050